CLINICAL TRIAL: NCT04393818
Title: A Double-blinded Randomized Controlled Trial to Examine the Effectiveness of a Mobile-based Intervention to Reduce Mental Health Problems in Healthcare Workers at the Frontline Against COVID-19 in Spain: the PsyCovidApp Trial
Brief Title: Mobile Phone Based Intervention to Protect Mental Health in Healthcare Workers at Frontline Against COVID19
Acronym: PsyCovid_App
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Collaborators: Universidad de las Islas Baleares (Unknown); Hospital Miguel Servet (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Andalusian School of Public Health (Other Government); Hospital Son Espases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: COVID-19/06
Record Dates: First submitted 2020-05-18; First posted 2020-05-19 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Mental Health Disorder; Depression; Posttraumatic Stress Disorder; Burnout; Anxiety Disorders
MeSH Terms: conditions — Mental Disorders; Depression; Stress Disorders, Post-Traumatic; Burnout, Psychological; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be blinded, as both the intervention and the control group will receive an App with information about management of mental health problems targeted at healthcare providers. The statisticians and outcome assessors (in this case the psychologists who will undertake the pre and post intervention psychological evaluations) will also be blinded. Only the PI and a research assistance will be unblinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention App (Experimental): Participants allocated to the intervention App will receive access to a fully operational mobile phone App. The App will be used to deliver psychoeducational materials (written and audio-visual), including: emotional training (mindfulness, moral harm, skills to manage emotions), lifestyles behaviour promotion (physical activity, diet, substance abuse, sleep), work environment, and social support.
  Interventions: Behavioral: Intervention App
- Control App (Sham Comparator): Participants allocated to the control App will receive access to a a fully operational mobile phone App with limited contents about management and prevention of mental health problems. Although this group will also receive psychoeducation, the content will be reduced to general, written recommendations.
  Interventions: Behavioral: Intervention App

INTERVENTIONS:
Behavioral: Intervention App — Participants allocated to the intervention App will receive access to a fully operational mobile phone App. The App will be used to deliver psychoeducational materials (written and audio-visual), including: emotional training (mindfulness, moral harm, skills to manage emotions), lifestyles behaviour promotion (physical activity, diet, substance abuse, sleep disorders), work environment, and social support.

SUMMARY:
This study aims at evaluating the effectiveness of a mobile phone based intervention to prevent and manage mental health problems in healthcare workers at the frontline against COVID-19 in Spain. The intervention will consist in psychoeducation, delivered via a mobile App. Participants will be followed up during two weeks. The primary outcome will be symptomatology of depression, anxiety or stress.

DETAILED DESCRIPTION:
Healthcare workers (HCWs) commonly present high levels of anxiety, depression, posttraumatic stress, acute disorder and burnout, both during and after viral outbreaks. Although educational and multifaceted interventions might mitigate the development of mental health problems, the certainty on the evidence is very low. The aim of this double-blinded randomized clinical trial is to examine the impact of a mobile phone based intervention to prevent and manage mental health problems in healthcare workers at the frontline against COVID-19 in Spain.

The trial will include HCWs having provided healthcare to patients with COVID19 in a healthcare centre (any setting) in Spain during the viral outbreak in Spain. Professionals from any medical speciality and role (doctors, nurses, nurse assistance, etc.) with access to a smartphone will be included. The investigators will collect expressions of interest via dissemination of the study through social media and key stakeholders (hospital managers, scientific societies and professional colleges). A team of psychologists will contact (via telephone) potential participants to confirm they meet the eligibility criteria (described above), obtain signed consent (audio-recorded), and carry out a psychological (pre-intervention) evaluation. The participants will then be randomly allocated to receive a fully functional App (full intervention) or an App with brief generic recommendations about mental health (control intervention). A post-intervention psychological assessment will be undertaken after two weeks. The primary outcome will be symptomatology of depression, anxiety or stress. Secondary outcomes will include posttraumatic stress, burnout, insomnia, and self-efficacy. After the two weeks follow-up, all participants allocated to the control intervention will be offered the full intervention.

ELIGIBILITY:
Inclusion Criteria:

Healthcare workers having provided healthcare to patients with COVID19 in a healthcare centre (any setting) during the viral outbreak in Spain.

We will include professionals from any medical speciality and role (doctors, nurses, nurse assistance, etc.).

Exclusion Criteria:

We will exclude healthcare workers not able to use, or with no access, to a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Depression, anxiety and stress | 2 weeks
  Depression, anxiety and stress scales (DASS21). Score range: 0 (worst outcome) to 21 (best outcome)

SECONDARY OUTCOMES:
Post-traumatic stress syndrome | 2 weeks
  Davidson Trauma Scale (DTS). The DTS is a 17-item, Likert-scale, self-report instrument that assesses the 17 DSM-IV symptoms of PTSD. Both a frequency and a severity score can be determined. The DTS yields a frequency score (ranging from 0 to 68), severity score (ranging from 0 to 68), and total score (ranging from 0 to 136). Higher scores are indicative a worse outcome.
Insomnia | 2 weeks
  Insomnia Severity Index. Score range: 0 (best outcome) to 28 (worst outcome)
Self Efficacy | 2 weeks
  General Self-Efficacy Scale. Score range: 10 (worst outcome) to 40 (best outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Ignacio Ricci-Cabello, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fiol-DeRoque MA, Serrano-Ripoll MJ, Jimenez R, Zamanillo-Campos R, Yanez-Juan AM, Bennasar-Veny M, Leiva A, Gervilla E, Garcia-Buades ME, Garcia-Toro M, Alonso-Coello P, Pastor-Moreno G, Ruiz-Perez I, Sitges C, Garcia-Campayo J, Llobera-Canaves J, Ricci-Cabello I. A Mobile Phone-Based Intervention to Reduce Mental Health Problems in Health Care Workers During the COVID-19 Pandemic (PsyCovidApp): Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 May 18;9(5):e27039. doi: 10.2196/27039. PMID 33909587
- [Derived] Serrano-Ripoll MJ, Ricci-Cabello I, Jimenez R, Zamanillo-Campos R, Yanez-Juan AM, Bennasar-Veny M, Sitges C, Gervilla E, Leiva A, Garcia-Campayo J, Garcia-Buades ME, Garcia-Toro M, Pastor-Moreno G, Ruiz-Perez I, Alonso-Coello P, Llobera J, Fiol-deRoque MA. Effect of a mobile-based intervention on mental health in frontline healthcare workers against COVID-19: Protocol for a randomized controlled trial. J Adv Nurs. 2021 Jun;77(6):2898-2907. doi: 10.1111/jan.14813. Epub 2021 Mar 6. PMID 33675247